CLINICAL TRIAL: NCT00555490
Title: Soy-Protein Intake, Cardio-Renal Indices and C-Reactive Protein in Type 2 Diabetes With Nephropathy: a 4-y Randomized Clincal Trial
Brief Title: Long-Term Effect of Soy Consumption on Cardio-Renal Indices and CRP in Type 2diabetes With Nephropathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IsfahanUMS
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2007-11-08 (Estimated); Status verified 2007-11

CONDITIONS: Kidney Transplantation
Keywords: Soy; Diabetes; Nephropathy
MeSH Terms: conditions — Diabetes Mellitus; Kidney Diseases | interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- 1 (Experimental)
  Interventions: Dietary Supplement: Soy protein

INTERVENTIONS:
Dietary Supplement: Soy protein — 35 % of protein from soy protein for 4-years

SUMMARY:
we conducted a longitudinal 4-year clinical trial to determine the long-term effects of soy consumption on lipid profiles, renal-function indices and CRP level among type 2 diabetic patients with nephropathy.

DETAILED DESCRIPTION:
Background: Several short-term trials on the effect of soy consumption on cardiovascular risks are available, but little evidence exists regarding the impact of long-term soy protein consumption among type 2 diabetic patients with nephropathy.

Objectives: To determine the effects of long-term soy consumption on cardiovascular risks, C-reactive protein and kidney-function indices among type 2 diabetic patients with nephropathy.

Design: This longitudinal randomized clinical trial was conducted among 41 type 2 diabetic patients with nephropathy (18 men and 23 women). Twenty patients in soy protein group consumed a diet containing 0.8 g protein/kg body weight (35% animal proteins, 35% textured soy protein, and 30% vegetable proteins) and 21 patients in control group consumed a similar diet containing 70% animal proteins and 30% vegetable proteins for 4-years.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes with Nephrophaty

Exclusion Criteria:

* Dialysis
* Transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2001-04; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
mortality or using dialysis | 4-years

CONTACTS AND LOCATIONS:
Overall Officials: Leila Azadbakht, PhD, Principal Investigator — Isfahan University of Medical Sciences, School of Health